CLINICAL TRIAL: NCT04990284
Title: A Randomized, Parallel Group, Multicentre, Multinational, Prospective, Open-label Exploratory Study to Evaluate the add-on Effect of Opicapone 50 mg or Levodopa 100 mg as First Strategy for the Treatment of Wearing-off in Patients With Parkinson's Disease.
Brief Title: eArly levoDopa With Opicapone in Parkinson's paTients wIth motOr fluctuatioNs.
Acronym: ADOPTION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067-403; 2020-002754-24 (EudraCT Number)
Record Dates: First submitted 2021-07-27; First posted 2021-08-04 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Adoption; Opicapone; Motor fluctuations
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone; Levodopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 50 mg opicapone once-daily (Experimental)
  Interventions: Drug: Opicapone
- 100 mg of L-DOPA (Experimental)
  Interventions: Drug: L-DOPA/DDCI

INTERVENTIONS:
Drug: Opicapone — 50 mg hard capsules. Oral administration, once-daily at bedtime, at least 1 hour before or after L-DOPA/carbidopa or benserazide (L-DOPA/DDCI).
  Other Names: BIA 9-1067
  Arms: 50 mg opicapone once-daily
Drug: L-DOPA/DDCI — L-DOPA/carbidopa or benserazide (L-DOPA/DDCI), 100/25 mg, oral administration
  Other Names: Levodopa
  Arms: 100 mg of L-DOPA

SUMMARY:
This is a randomized, parallel group, multicentre, multinational, prospective, open-label exploratory study in Parkinson's disease (PD) patients to evaluate the add-on efficacy of opicapone 50 mg or an extra dose of levodopa (L-DOPA) 100 mg as first strategy for the treatment of wearing-off.

DETAILED DESCRIPTION:
The study consists of a one-week screening period, four weeks of open-label treatment and two weeks of post-study follow-up. The total study duration for each patient will be approximately 7 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an informed consent form and to comply with all aspects of the study.
2. Male or female patients aged 30 years or older.
3. Diagnosed with idiopathic PD according to the UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria (2006) or according to the Movement Disorder Society (MDS) Clinical Diagnostic Criteria (2015).
4. Disease severity Stages I-III (Hoehn & Yahr staging) at ON.
5. Treated on a stable regimen for at least four weeks before screening with immediate-release L-DOPA/DDCI, three to four intakes per day, and up to maximum daily dose of 600 mg L-DOPA.
6. In case of any other anti-PD-treatments, they should be on a stable regimen for at least four weeks before screening, and not likely to need any adjustment during the study.
7. Signs of wearing-off phenomenon with average total daily OFF-time while awake of at least 1 hour, including the early morning pre-first dose OFF (i.e. the time between wake-up and response to the first L DOPA/DDCI dosage), despite optimal anti-PD therapy (based on Investigator's assessment).
8. Experiencing wearing-off phenomenon for at least 4 weeks but less than 2 years prior to screening.
9. For females: Postmenopausal for at least 2 years before screening, surgically sterile for at least 6 months before screening, or practicing effective contraception until the post-study visit. Female patients who request to continue with oral contraceptives must be willing to use non-hormonal methods of contraception in addition during the course of this study.
10. Have filled-in self-rating diary charts in accordance with the diary chart instructions and with ≤3 errors per day while awake, in the three consecutive days preceding randomization.
11. With at least 1 hour at OFF state per day, including the early morning pre-first dose OFF period (i.e. the time between wake-up and response to the first L DOPA/DDCI dosage), as recorded in at least two of the three-day self-rating diary charts for the three days preceding randomization.
12. Adequate compliance to relevant concomitant medication during the period between V1 and V2 (based on the Investigator's judgment).

Exclusion Criteria:

1. Non-idiopathic PD (atypical parkinsonism, secondary [acquired or symptomatic] parkinsonism, Parkinson-plus syndrome).
2. Severe and/or unpredictable OFF periods, according to Investigator's judgment.
3. Average total daily OFF-time while awake of >5 hours, including the early morning pre-first dose OFF, despite optimal anti-PD therapy (based on Investigator's assessment).
4. Treatment with prohibited medication: entacapone, tolcapone, monoamine oxidase (MAO) inhibitors (except selegiline up to 10 mg/day in oral formulation or 1.25 mg/day in buccal absorption formulation, rasagiline up to 1 mg/day or safinamide up to 100 mg/day), apomorphine or antiemetics with antidopaminergic action (except domperidone) within the last 4 weeks before screening.
5. Previous or planned (during the entire study duration) deep brain stimulation or stereotactic surgery (e.g. pallidotomy, thalamotomy).
6. Previous or current use of opicapone or L-DOPA/carbidopa intestinal gel infusion.
7. Use of any other investigational product (IP), currently or within the 3 months (or within 5 half-lives of the IP, whichever is longer) before screening.
8. Past (within the past year) or present history of suicidal ideation or suicide attempts.
9. Current or previous (within the past year) alcohol or substance abuse excluding caffeine or nicotine.
10. Phaeochromocytoma, paraganglioma, or other catecholamine secreting neoplasms.
11. Known hypersensitivity to the excipients of IP (including lactose intolerance, galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption).
12. History of neuroleptic malignant syndrome or non-traumatic rhabdomyolysis.
13. History of severe hepatic impairment (Child-Pugh Class C).
14. Current or previous (within the past year) diagnosis of psychosis, severe major depression or other psychiatric disorders that, based on the Investigator's judgment, might place the patient at increased risk or interfere with assessments.
15. Any medical condition that might place the patient at increased risk or interfere with assessments.
16. For females: Pregnant or breastfeeding.
17. Employees of the Investigator, study centre, Sponsor, clinical research organisation and study consultants, when employees are directly involved in this study or other studies under the direction of this Investigator or study centre, and their family members.
18. Persons committed to an institution by virtue of an order issued either by the judicial or other authorities.
19. With an average total daily OFF-time while awake of >5 hours, including the early morning pre-first dose OFF period (i.e. the time between wake-up and response to the first L DOPA/DDCI dosage), as recorded in at least two of the three-day self-rating diary charts for the three days preceding randomization

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Change in Absolute OFF-time from baseline to end of study | up to 7 weeks
  OFF = Time when medication has worn off and is no longer providing benefit with regard to mobility, slowness, and stiffness.
Proportion of patients with one hour or more reduction in Absolute OFF-time from baseline to end of study (OFF-time responders) | up to 7 weeks
  OFF = Time when medication has worn off and is no longer providing benefit with regard to mobility, slowness, and stiffness.
Change in Absolute ON-time from baseline to end of study | up to 7 weeks
  ON = Time when medication is providing benefit with regard to mobility, slowness, and stiffness.
Proportion of patients with one hour or more increase in Absolute ON-time from baseline to end of study (ON-time responders) | up to 7 weeks
  ON = Time when medication is providing benefit with regard to mobility, slowness, and stiffness.
Change in Percentage OFF-time between baseline and end of study | up to 7 weeks
  OFF = Time when medication has worn off and is no longer providing benefit with regard
Change in Percentage ON-time between baseline and end of study | up to 7 weeks
  ON = Time when medication is providing benefit with regard to mobility, slowness, and stiffness.

CONTACTS AND LOCATIONS:
Locations (25):
- Germany (8):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Parkinson-Klinik Ortenau GmbH&Co KG, Wolfach, Baden-Wurttemberg
  - Klinik Haag i. OB, Haag in Oberbayern, Bavaria
  - Universitaetsklinikum Wuerzburg, Würzburg, Bavaria
  - Praxis Dr. Oehlwein, Gera, Thuringia
  - Asklepios Fachklinikum Stadtroda, Stadtroda, Thuringia
  - Charite Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Praxis Dr. med. Kirsten Hahn, Berlin
- Italy (4):
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria- Università degli Studi della Campania "Luigi Vanvitelli", Napoli
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliera Santa Maria di Terni, Terni
- Portugal (2):
  - Hospital Beatriz Ângelo, Loures, Lisbon District
  - CNS-Campus Neurologico Senior, Torres Vedras, Lisbon District
- Spain (7):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital de Sant Joan Despi Moises Broggi, Sant Joan Despí, Barcelona
  - Complejo Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Ruber Internacional, Madrid
  - Complejo Hospitalario Universitario de Orense, Ourense
- United Kingdom (4):
  - Royal Devon and Exeter Hospital (Wonford), Exeter, Devon
  - University Hospitals Plymouth, Plymouth, Devon
  - King's College Hospital, London, Greater London
  - Newcastle University- Clinical Ageing Research Unit, Newcastle upon Tyne, Tyne & Wear

IPD SHARING:
Plan to Share IPD: No